CLINICAL TRIAL: NCT02457624
Title: A Prospective Cohort Study for Development of Korean Gastric Cancer Prediction Model and Tailored Gastric Cancer Screening Program
Brief Title: Gastric Cancer Screening Quality Improvement System Establishment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Su Jin Chung, Associated Professor, Seoul National University Hospital
Other Study IDs: 1503-044-655
Record Dates: First submitted 2015-03-25; First posted 2015-05-29 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Gastric Cancer; Gastritis, Atrophic; Intestinal Metaplasia
Keywords: gastric cancer; chronic atrophic gastritis; intestinal metaplasia
MeSH Terms: conditions — Stomach Neoplasms; Gastritis, Atrophic | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Experienced endoscopists: All the experienced endoscopists will receive education and feedback on the diagnosis for premalignant lesion of chronic atrophic gastritis and intestinal metaplasia
  Interventions: Behavioral: Education and feedback

INTERVENTIONS:
Behavioral: Education and feedback — Experienced endoscopists will receive education on Kimura-Takemoto classification and feedback for their answers for classification tests.

SUMMARY:
Experienced endoscopists will perform endoscopy during the study period and the detection rate of gastric premalignant lesion, correlation between endoscopic and serologic diagnosis of premalignant lesions and inter-observer agreement rate will be analyzed before and after the education.

DETAILED DESCRIPTION:
This study is an extension of quality assurance program in Seoul National University Hospital Healthcare System Gangnam Center. This study is composed of four periods. First, the detection rate of gastric premalignant lesions and the correlation between endoscopic and serologic diagnosis of premalignant lesions will be analyzed retrospectively from March 2008 till February 2009 and from March 2013 till February 2014, when the levels of serum pepsinogen were achieved from the patients. In the second period from March 2015 till April 2015, quality assurance program will be activated. Endoscopists will be educated on the Kimura-Takemoto classification for chronic atrophic gastritis. After that their diagnosis will be tested and they will have feedback and discussion all together. In this period, inter-observer agreement rate will be assessed serially. Third, prospective trial will run from May 2015 till April 2020, in which all the endoscopists' detection rate of gastric premalignant lesion, the correlation between endoscopic and serologic diagnosis of premalignant lesions, and their inter-observer agreement will be analyzed. Finally, cumulative incidence and mortality rate of gastric cancer and incidence rate of gastric dysplasia will be investigated until December 2020.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received endoscopy in Seoul National University Hospital Healthcare System Gangnam Center from 2008 till 2020.

Exclusion Criteria:

* Age < 18 years
* Those who refused to be included in the research
* History of gastric cancer
* Current medication with proton pump inhibitor, non-steroidal anti-inflammatory drug or aspirin
* Active/healing stage of gastric ulcer or gastric ulcer scar
* Active/healing stage of duodenal ulcer
* History of previous surgical or endoscopic resection of stomach

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who received colonoscopy in Seoul National University Hospital Healthcare System Gangnam Center from 2008 till 2020.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Estimated)
Dates: Start 2008-03; Primary Completion 2020-04 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Detection rate for gastric premalignant lesion | 7 years

SECONDARY OUTCOMES:
Correlation between endoscopic and serologic diagnosis of premalignant lesions | 7 years
Inter-observer agreement rate for the diagnosis of premalignant lesions | 2 months
Detection rate for gastric cancer | 7 years
Detection rate for gastric dysplasia | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Su Jin Chung, MD.PhD., Principal Investigator — Department of Internal Medicine and Healthcare Research Institute, Healthcare System Gangnam Center, Seoul National University Hospital
Locations (1):
- Healthcare System Gangnam Center, Seoul National University Hospital, Seoul, South Korea